CLINICAL TRIAL: NCT02797210
Title: Efficacy of Orbital Frontal Cortex Repetitive Transcranial Magnetic Stimulation Magnetic Stimulation in the Treatment of Refractory Depression
Brief Title: Examining the Efficacy of Orbitofrontal Cortex rTMS for Depression
Acronym: OFC-rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-5094
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2016-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham then Active Stimulation (Experimental): Sham repetitive transcranial magnetic stimulation (rTMS) to right orbitofrontal cortex, twice daily, 5 days per week for 3 weeks, then active rTMS to right orbitofrontal cortex, twice daily, 5 days per week for 3 weeks
  Interventions: Device: Continuous theta-burst stimulation
- Active then Sham Stimulation (Experimental): Active repetitive transcranial magnetic stimulation (rTMS) to right orbitofrontal cortex, twice daily, 5 days per week for 3 weeks, then sham rTMS to right orbitofrontal cortex, twice daily, 5 days per week for 3 weeks
  Interventions: Device: Continuous theta-burst stimulation

INTERVENTIONS:
Device: Continuous theta-burst stimulation

SUMMARY:
This trial will compare the efficacy of active inhibitory OFC-rTMS to sham OFC-rTMS in major depression. The trial will include structural and functional MRI, EEG, and behavioral measures obtained before, during, and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. are outpatients
2. are voluntary and competent to consent to treatment
3. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of major depressive disorder (MDD), single or recurrent
4. are between the ages of 18 and 65
5. have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of > 3 in the current
6. have a score > 18 on the HAMD-17
7. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
8. able to adhere to the treatment schedule
9. Pass the TMS adult safety-screening (TASS) questionnaire
10. have normal thyroid functioning based on pre-study blood work.

Exclusion Criteria:

1. have a MINI-International Neuropsychiatric (MINI) confirmed diagnosis of substance dependence or abuse within the last 3 months
2. have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
3. have active suicidal intent
4. are pregnant
5. have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
6. have a MINI diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, assessed by a study investigator to be primary and causing greater impairment than MDD
7. have a diagnosis of any personality disorder, and assessed by a study investigator to be primary and causing greater impairment than MDD
8. have failed a course of electroconvulsive therapy (ECT) in the current episode or previous episode
9. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
10. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
11. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
12. clinically significant laboratory abnormality, in the opinion of the study investigator
13. currently (or in the last 4 weeks) take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
14. non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
17-Item Hamilton Rating Scale for Depression (HAMD-17) | Baseline, after each week of treatment (i.e. after 5 days of treatment) and at 1, 4, and 12 weeks post-treatment.
  Outcome measured by a change in HAMD-17 score from baseline to 2 weeks post-treatment. A 50% improvement in the score is considered a response to rTMS. A final score of <8 is categorized as remission.

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Daily for 6 weeks

OTHER OUTCOMES:
Magnetic Resonance Imaging (MRI) | 1 week pre- and 1 week post-treatment
  10 min resting-state functional MRI (rs-fMRI) at 3 Tesla (3T)
Electroencephalography (EEG) | Day 1 (First day of treatment), Day 15, and Day 30 (Final day of treatment)]
  10 min resting-state and task-based (response inhibition, reward sensitivity) acquisitions

CONTACTS AND LOCATIONS:
Locations (1):
- UHN MRI-Guided rTMS Clinic, Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No